CLINICAL TRIAL: NCT00220298
Title: Open One-arm Study to Investigate Safety and Efficacy of Intramuscular Injections of 1000 mg Testosterone Undecanoate (TU) in Hypogonadal Men at Variable Intervals During a 136-week to 192-week Treatment Including Pharmacokinetics
Brief Title: Assessment of Long Term Treatment With Testosterone Undecanoate in Males With Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91186; 306605 (Other: company internal)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Testosterone undecanoate (TU) - NebidoTM

INTERVENTIONS:
Drug: Testosterone undecanoate (TU) - NebidoTM — Drug treatment with 14 injections of one ampoule of Nebido (1000 mg of testosterone undecanoate) at individually adjusted injection intervals

SUMMARY:
This study will evaluate the preparation of testosterone undecanoate under conditions which resemble real-life situations.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadal men, aged 18-75 years with low serum total testosterone (TT) levels and symptoms of androgen deficiency

Exclusion Criteria:

* Tumors of the prostate or the male mammary gland including suspicion thereof. Past or present liver tumors or chronic hepatic disease with impairment of liver function, Severe acne.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2003-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of long term treatment with TU under real-life conditions | Every 3 months during treatment and after final injection

SECONDARY OUTCOMES:
Assessment of treatment satisfaction by patient | 6,10, and 14 injections

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- Germany (12):
  - Nuremberg, Bavaria
  - Marburg, Hesse
  - Wolfsburg, Lower Saxony
  - Münster, North Rhine-Westphalia
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Naumburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Eisenberg, Thuringia
  - Gera, Thuringia
  - Jena, Thuringia
  - Leipzig

REFERENCES:
- [Result] Behre HM and Elliesen J. Safety and efficacy of intramuscular injections of 1000 mg testosterone undecanoate: A prospective multicenter study in hypogonadal men under conditions resembling real-life situations. Proceedings of the 22nd Annual European Association of Urology (EAU); 2007 Mar 22; Berlin, Germany. Eur Urol Suppl 2007;6(2):108.